CLINICAL TRIAL: NCT00811083
Title: DMSA Treatment of Children With Autism and Heavy Metal Toxicity
Brief Title: Dimercaptosuccinic Acid (DMSA) Treatment of Children With Autism and Heavy Metal Toxicity
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Southwest College of Naturopathic Medicine (Other)
Responsible Party: Matthew Baral and James B. Adams, Southwest College of Naturopathic Medicine
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: DMSA
Record Dates: First submitted 2008-12-17; First posted 2008-12-18 (Estimated); Last update posted 2008-12-18 (Estimated); Status verified 2008-12

CONDITIONS: Autism
Keywords: autism; toxic metals; DMSA; dimercaptosuccinic acid; chelation
MeSH Terms: conditions — Autistic Disorder | interventions — Succimer

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- DMSA- 1 round (Active Comparator): Subjects receive 1 round of DMSA (10 mg/kg-dose, 9 doses over 3 days), followed by 3 months of placebo
  Interventions: Drug: DMSA - dimercaptosuccinic acid
- DMSA-7 rounds (Active Comparator): Participants receive 7 rounds of DMSA over 4 months; each round consists of 3 days of DMSA (10 mg/kg-dose, 9 doses over 3 days), followed by 11 days off (no treatment), and then repeating.
  Interventions: Drug: DMSA - dimercaptosuccinic acid

INTERVENTIONS:
Drug: DMSA - dimercaptosuccinic acid — dose of 10 mg/kg bodyweight 3 doses/day, for 3 days, followed by 11 days off
  Other Names: Succimer

SUMMARY:
Many children with autism have a reduced level of glutathione and a reduced ability to excrete mercury, resulting in elevated levels in their bodies as demonstrated by blood, hair, provoked urine, and baby tooth testing. Our earlier studies have demonstrated that DMSA, an FDA-approved medication for treating lead poisoning in children, is effective in increasing excretion of mercury and other toxic metals. Based on many clinical reports, we hypothesize that a 3-month treatment with glutathione and DMSA will result in a reduction of autistic symptoms in some children with autism.

DETAILED DESCRIPTION:
This study will assess the safety and efficacy of the use of DMSA (an FDA-approved medication for treating lead poisoning in children) for the off-label treatment of symptoms of autism in children with autism and significant body burden of toxic metals.

ELIGIBILITY:
Inclusion Criteria:

Phase One

1. Children with autism spectrum disorder
2. Age 3-8 years (up to the day before the ninth birthday).
3. At least a two-month history of taking a multi-vitamin/mineral supplement with at least the RDA of zinc, and continuing to take that during Phase One and Two.

Phase Two:

1. Excretion of high amounts of toxic metals in phase one
2. Normal kidney/liver function, serum transaminases, and Complete Blood Count (CBC) (based on a blood test which will be conducted as part of Phase Two)
3. No changes in medication, supplements, diet, or behavioral interventions during the study

Exclusion Criteria:

Phase One and Two:

* No mercury amalgam dental fillings.
* No previous use of DMSA or other prescription chelators (except for 1-time challenges).
* No anemia or currently being treated for anemia due to low iron.
* No known allergies to DMSA
* No liver or kidney disease

Ages: 3 Years to 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 80 (Actual)
Dates: Start 2005-05; Primary Completion 2007-04 (Actual); Study Completion 2007-04 (Actual)

PRIMARY OUTCOMES:
Determine the effect of DMSA therapy on the symptoms of autism | 4 month
Determine the safety of DMSA therapy by pre/post assessment of complete blood count, standard chem panel including liver/kidney function, and excretion of essential minerals | 4 months

SECONDARY OUTCOMES:
Determine if the initial severity of autism correlates with the excretion of toxic metals | 1 month

CONTACTS AND LOCATIONS:
Overall Officials: James B. Adams, PhD, Principal Investigator — Southwest College of Naturopathic Medicine; Matthew Baral, ND, Principal Investigator — Southwest College of Naturopathic Medicine
Locations (1):
- Southwest College of Naturopathic Medicine, Tempe, Arizona, United States